CLINICAL TRIAL: NCT06800807
Title: Metacognitive Beliefs and Eating and Nutrition Disorders in Adolescents With Eating and Nutrition Disorders
Brief Title: Metacognitive Beliefs in Adolescents With Eating and Nutrition Disorders
Acronym: METAED
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C412
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Feeding and Eating Disorders
Keywords: metabeliefs; metacognition; brooding; rumination; anorexia nervosa; bulimia nervosa; binge eating disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Rumination Syndrome; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder | interventions — Eating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eating and nutrition disorders (END): Female patients aged between 12 and 17 years, of Italian nationality, who present a diagnosis relating to the END framework according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
  Interventions: Other: Observation of several factors involved in eating and nutrition disorders
- Control group: Female subjects of the same age and of Italian nationality, belonging to the general population.
  Interventions: Other: Observation of several factors involved in eating and nutrition disorders

INTERVENTIONS:
Other: Observation of several factors involved in eating and nutrition disorders — Observation of symptomatology of eating and nutrition disorders, metacognitive beliefs, brooding and rumination.

SUMMARY:
The present study aims to study the presence of metacognitive beliefs in adolescent subjects with eating and nutrition disorders (END) compared with a control group composed of subjects of the same sex and age belonging to the general population.

ELIGIBILITY:
Eating and nutrition disorders (END)

Inclusion Criteria:

* Female sex
* Age: 12 to 17 years
* Italian nationality
* Diagnosis relating to the END framework according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).

Exclusion Criteria:

* Absence of signed Informed Consent

Control group

Inclusion Criteria:

* Female sex
* Age: 12 to 17 years
* Italian nationality

Exclusion Criteria:

* Absence of signed Informed Consent

Ages: 12 Years to 17 Years | Sex: Female
Age Groups: Child
Study Population: 36 patients aged between 12 and 17 years, females, of Italian nationality, who present a diagnosis relating to the END framework according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
  These patients will be compared with a control group made up of 36 subjects of the same sex, age, and nationality, belonging to the general population.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Metacognitive beliefs | Baseline
  Metacognition Questionnaire (MCQ-30; Cartwright-Hatton & Wells, 1997), a self-report test composed of 30 items on a 4-point Likert scale from 1 (I do not agree) to 4 (I completely agree 'agreement)
Brooding | Baseline
  Penn State Worry Questionnaire (PSWQ; Meyer et at., 1990), a self-report test composed of 16 items on a 5-point Likert scale from 1 (not at all typical) to 5 (very typical)
Rumination | Baseline
  Ruminative Response Scale (RRS; Nolen-Hoeksema and Morrow, 1991), a self-report test composed of 20 items on a 4-point Likert scale from 1 (almost never) to 4 (almost always)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy